CLINICAL TRIAL: NCT00838552
Title: Prospective Analysis of Markers of Airway Inflammation and Remodeling in Bronchoalveolar Lavage Fluid From Children With Asthma.
Brief Title: Markers of Airway Inflammation in BAL Fluid From Children With Asthma
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NJ HS-2178
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Asthma
Keywords: asthma inflammation bronchoscopy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 Asthma subjects: Children with asthma undergoing clinically indicated bronchoscopy at National Jewish Health.
- 2 Non-asthma subjects: Children with other respiratory diseases than asthma undergoing clinically indicated bronchoscopy at National Jewish Health.

SUMMARY:
The study compares the biochemical markers in bronchoalveolar lavage samples from asthmatic children to those markers found in non-asthmatic children with other respiratory diseases. The investigators hypothesize that certain markers will be associated specifically with asthma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or younger
* Scheduled for bronchoscopy at National Jewish Health for persistent asthma, persistent, poorly controlled wheezing, chronic cough, GERD, atelectasis, bronchopulmonary dysplasia, infection.
* Consent and assent from parent and patient [if appropriate].

Exclusion Criteria:

* Unwillingness to consent/assent to retrieval of BAL fluid for research analysis.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients undergoing bronchoscopy at National Jewish Health
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2007-10; Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
The measurement of levels of lipopolysaccharides [LPS], which mediates airway inflammation, in bronchoalveolar lavage [BAL] fluid from children with asthma and comparison to LPS levels in children with non-asthma respiratory diseases | Single time point

SECONDARY OUTCOMES:
Characterization of the inflammatory cytokine and chemokine profiles in bronchoalveolar lavage [BAL] fluid in children with asthma and comparison to the profile for children with non-asthma respiratory diseases. | Single time point

CONTACTS AND LOCATIONS:
Overall Officials: Pia Hauk, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] Wenzel SE, Fowler AA 3rd, Schwartz LB. Activation of pulmonary mast cells by bronchoalveolar allergen challenge. In vivo release of histamine and tryptase in atopic subjects with and without asthma. Am Rev Respir Dis. 1988 May;137(5):1002-8. doi: 10.1164/ajrccm/137.5.1002. PMID 2461667
- [Background] Bousquet J, Chanez P, Lacoste JY, Barneon G, Ghavanian N, Enander I, Venge P, Ahlstedt S, Simony-Lafontaine J, Godard P, et al. Eosinophilic inflammation in asthma. N Engl J Med. 1990 Oct 11;323(15):1033-9. doi: 10.1056/NEJM199010113231505. PMID 2215562
- [Background] Vignola AM, Chanez P, Chiappara G, Siena L, Merendino A, Reina C, Gagliardo R, Profita M, Bousquet J, Bonsignore G. Evaluation of apoptosis of eosinophils, macrophages, and T lymphocytes in mucosal biopsy specimens of patients with asthma and chronic bronchitis. J Allergy Clin Immunol. 1999 Apr;103(4):563-73. doi: 10.1016/s0091-6749(99)70225-3. PMID 10200002
- [Background] Woodman L, Sutcliffe A, Kaur D, Berry M, Bradding P, Pavord ID, Brightling CE. Chemokine concentrations and mast cell chemotactic activity in BAL fluid in patients with eosinophilic bronchitis and asthma, and in normal control subjects. Chest. 2006 Aug;130(2):371-8. doi: 10.1378/chest.130.2.371. PMID 16899834
- [Background] Krawiec ME, Westcott JY, Chu HW, Balzar S, Trudeau JB, Schwartz LB, Wenzel SE. Persistent wheezing in very young children is associated with lower respiratory inflammation. Am J Respir Crit Care Med. 2001 May;163(6):1338-43. doi: 10.1164/ajrccm.163.6.2005116. PMID 11371398